CLINICAL TRIAL: NCT03573544
Title: A Phase I/II, Open-Label, Dose Escalation and Cohort Expansion Study Evaluating the Safety, Pharmacokinetics (PK), Pharmacodynamics (PD), and Therapeutic Activity of OBI-888 in Patients With Locally Advanced or Metastatic Solid Tumors.
Brief Title: This Study is to Evaluate Safe and Effective Treatment Dose of OBI-888 in Patients With Locally Advanced or Metastatic Solid Tumors.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: OBI-888 no longer fulfills our goal of developing cost-effective therapies for cancer patients
Sponsor: OBI Pharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OBI-888-001
Record Dates: First submitted 2018-05-07; First posted 2018-06-29 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Solid Tumors; Locally Advanced Solid Tumors
Keywords: mAbs; monoclonal antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- OBI-888 Escalation Phase (Experimental): Part A: Three cohorts of escalating dose levels of OBI-888 5, 10, and 20 mg/kg liquid form for intravenous infusion to establish maximum tolerated dose (MTD).
  Interventions: Drug: OBI-888; Device: Globo H IHC Assay
- OBI-888 Expansion Phase (Experimental): Part B: Five cohorts at dose level 20 mg/kg of liquid form OBI-888 for intravenous infusion.
  Interventions: Drug: OBI-888; Device: Globo H IHC Assay

INTERVENTIONS:
Drug: OBI-888 — For the dose-escalation phase, OBI-888 will be given weekly at the dose levels of 5, 10, and 20 mg/kg.
  Arms: OBI-888 Escalation Phase
Drug: OBI-888 — For the dose-expansion phase, OBI-888 will be given weekly at 20 mg/kg dose level.
  Arms: OBI-888 Expansion Phase
Device: Globo H IHC Assay — This assay will be used to identify eligible patients who may clinically benefit from the OBI-888 treatment, defined by Globo H expression.

SUMMARY:
The purpose of this study is to establish the maximum tolerated dose (MTD) of OBI-888 as monotherapy. And to characterize the safety and preliminary clinical activity profile of the MTD dose of OBI-888 administered as monotherapy in patients with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria in order to be included in the study:

1. Male or female patients, 18 years of age or older at the time of consent.
2. Provide written informed consent prior to performing any study-related procedure.
3. Histologically or cytologically confirmed patients with advanced or metastatic solid tumors for both Dose Escalation and Expansion cohort.
4. Patients must have been treated with established standard-of-care therapy, or physicians have determined that such established therapy is not sufficiently efficacious, or patients have declined to receive standard-of-care therapy.
5. Measurable disease (i.e., at least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Adequate organ function defined as:

   * Hepatic:

     * Serum alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN), ≤5 × ULN in the presence of liver metastases
     * Serum aspartate aminotransferase (AST) ≤3 × ULN, ≤5 × ULN in presence of liver metastases
     * Serum bilirubin ≤1.5 × ULN
   * Renal:

     * Creatinine clearance >30 mL/minute using Cockcroft Gault equation
   * Hematologic:

     * Absolute neutrophil count ≥1000/µL
     * Platelets ≥75,000/µL
     * Hemoglobin ≥8 g/dL
8. Patient is willing and able to comply with all protocol required assessments, visits, and procedures, including pretreatment tumor biopsy. Archival tumor biopsies are acceptable at baseline.
9. Females of childbearing potential must have negative urine or serum pregnancy test prior to starting study therapy, and agree to use a reliable form of contraceptive during the study treatment period and for at least 120 days following the last dose of study drug.

   Subject not of childbearing potential (i.e., permanently sterilized, postmenopausal) can be included in study. Postmenopausal is defined as 12 months with no menses without an alternative medical cause.

   Male patients must agree to use an adequate method of contraception during the study treatment period and for at least 120 days following the last dose of study drug.
10. Cannot be breast feeding.
11. Patients in Part B (Cohort expansion); must have a qualifying, documented Globo H H-score in sponsor-selected tumor types to be enrolled in the respective cohort:

    * Cohort 1: Pancreatic cancer
    * Cohort 2: Esophageal cancer
    * Cohort 3: Gastric cancer
    * Cohort 4: Colorectal cancer
    * Cohort 5: Basket (any solid tumor type other than those included in Cohorts 1 through 4)

Exclusion Criteria:

Patients meeting any of the following criteria are ineligible to participate in this study:

1. Less than 3 weeks, from prior cytotoxic chemotherapy or radiation therapy; and less than 5 half-lives or 3 weeks from biological therapies, whichever is shorter, prior to the first dose of OBI-888.
2. Has undergone a major surgical procedure (as defined by the investigator) or significant traumatic injury within 28 days prior to the first dose of OBI-888.
3. Presence of an active autoimmune or inflammatory disease requiring systemic treatment within the past 2 months or a documented history of clinically severe autoimmune disease that requires systemic steroids or other immunosuppressive medications. Local steroid injections, intermittent use of topical, inhaled, ophthalmologic, intra-articular, topical, or intranasal corticosteroids, or systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent would not be excluded from the study.
4. Presence of primary immunodeficiency or receiving systemic steroids of >10 mg/day of prednisone or equivalent or other immunosuppressive agents within 14 days prior to the first dose of OBI 888.
5. Has active bacterial, viral, fungal, or mycobacterial infection requiring systemic therapy, including known infection with human immunodeficiency virus (HIV) or active infection with hepatitis B virus or hepatitis C virus.
6. Patients with a history of solid organ transplant.
7. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to Grade 0 or 1 (using National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.03), except for alopecia and laboratory values listed in the inclusion criteria.
8. Receipt of any prior therapy targeting Globo H.
9. Known hypersensitivity to OBI 888 or its excipients.
10. Has known, untreated central nervous system metastases and/or leptomeningeal metastases.
11. Any medical co morbidity or psychiatric illness that is life threatening or, in the opinion of the Investigator, renders the patient unsuitable for participation in a clinical trial due to possible noncompliance, would place the patient at an unacceptable risk and/or potential to affect interpretation of results of the study.
12. Is receiving any concurrent prohibited medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia Tsimberidou, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (9):
- United States (6):
  - Scripps Clinic Torrey Pines, La Jolla, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - West Cancer Center and Research Institute, Germantown, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, Dose Escalation - OBI-888 5 mg/kg: OBI-888 5 mg/kg was administered as an IV infusion for approximately 90 minutes (±10 minutes) on Days 1, 8, 15 and 22 of each 28-day cycle for 2 cycles
- Part A, Dose Escalation - OBI-888 10 mg/kg: OBI-888 10 mg/kg was administered as an IV infusion for approximately 90 minutes (±10 minutes) on Days 1, 8, 15 and 22 of each 28-day cycle for 2 cycles
- Part A, Dose Escalation - OBI-888 20 mg/kg; Part B, Cohort Expansion - Cohort 1, Pancreatic; Part B, Cohort Expansion - Cohort 2, Esophageal; Part B, Cohort Expansion - Cohort 3, Gastric; Part B, Cohort Expansion - Cohort 4, Colorectal; Part B, Cohort Expansion - Cohort 5, Basket: OBI-888 20 mg/kg was administered as an IV infusion for approximately 90 minutes (±10 minutes) on Days 1, 8, 15 and 22 of each 28-day cycle for 2 cycles
Period: Overall Study
Arm/Group | Part A, Dose Escalation - OBI-888 5 mg/kg | Part A, Dose Escalation - OBI-888 10 mg/kg | Part A, Dose Escalation - OBI-888 20 mg/kg | Part B, Cohort Expansion - Cohort 1, Pancreatic | Part B, Cohort Expansion - Cohort 2, Esophageal | Part B, Cohort Expansion - Cohort 3, Gastric | Part B, Cohort Expansion - Cohort 4, Colorectal | Part B, Cohort Expansion - Cohort 5, Basket
Started | 5 | 3 | 6 | 8 | 7 | 8 | 9 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 3 | 6 | 8 | 7 | 8 | 9 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Not completed — Disease progression | 3 | 3 | 6 | 4 | 5 | 7 | 6 | 7

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all enrolled subjects who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Dose Escalation - OBI-888 5 mg/kg | Part A, Dose Escalation - OBI-888 10 mg/kg | Part A, Dose Escalation - OBI-888 20 mg/kg | Part B, Cohort Expansion - Cohort 1, Pancreatic | Part B, Cohort Expansion - Cohort 2, Esophageal | Part B, Cohort Expansion - Cohort 3, Gastric | Part B, Cohort Expansion - Cohort 4, Colorectal | Part B, Cohort Expansion - Cohort 5, Basket | Total
Number analyzed (Participants) | 5 | 3 | 6 | 8 | 7 | 8 | 9 | 8 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12.86) | 57.7 (9.45) | 64.5 (12.1) | 63.8 (13.29) | 57.4 (9.36) | 64.9 (9.69) | 52.9 (14.84) | 60.6 (8.07) | 59.8 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 3 | 6 | 0 | 3 | 2 | 5 | 27
  Male | 0 | 0 | 3 | 2 | 7 | 5 | 7 | 3 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 3 | 6 | 7 | 0 | 4 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 3 | 1 | 5 | 5 | 1 | 1 | 9 | 4 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity (NIH/OMB): Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Ethnicity (NIH/OMB): Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ethnicity (NIH/OMB): East Asian | 0 | 0 | 0 | 3 | 6 | 7 | 0 | 3 | 19
  Ethnicity (NIH/OMB): Other | 2 | 2 | 3 | 4 | 1 | 1 | 8 | 3 | 24
  Ethnicity (NIH/OMB): Unknown or not reported | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CR, PR, SD) (%)
Description: Assessment of OBI-888 clinical benefit rate for dose escalation and cohort expansion phases of the OBI-888-001 study.
Time Frame: Every 8 weeks (±1 week) for 6 months, then every 12 weeks (±1 week) until progression or off-study criteria, up to 1 year.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Part A, Dose Escalation - OBI-888 5 mg/kg | Part A, Dose Escalation - OBI-888 10 mg/kg | Part A, Dose Escalation - OBI-888 20 mg/kg | Part B, Cohort Expansion - Cohort 1, Pancreatic | Part B, Cohort Expansion - Cohort 2, Esophageal | Part B, Cohort Expansion - Cohort 3, Gastric | Part B, Cohort Expansion - Cohort 4, Colorectal | Part B, Cohort Expansion - Cohort 5, Basket
Number analyzed (Participants) | 5 | 3 | 6 | 8 | 7 | 8 | 9 | 8
Percentage | 20 [0.5 to 71.6] | 66.7 [9.4 to 99.2] | 16.7 [0.4 to 64.1] | 12.5 [0.3 to 52.7] | 14.3 [0.4 to 57.9] | 25 [3.2 to 65.1] | 22.2 [2.8 to 60.0] | 25 [3.2 to 65.1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through 12 months
Description: Treatment-emergent adverse events (TEAEs) in Parts A or B experienced by ≥5% of total subjects in Part A and Part B. TEAEs are presented by decreasing incidence for the total of subjects in Part A and Part B
Arm/Group | Part A, Dose Escalation - OBI-888 5 mg/kg | Part A, Dose Escalation - OBI-888 10 mg/kg | Part A, Dose Escalation - OBI-888 20 mg/kg | Part B, Cohort Expansion - Cohort 1, Pancreatic | Part B, Cohort Expansion - Cohort 2, Esophageal | Part B, Cohort Expansion - Cohort 3, Gastric | Part B, Cohort Expansion - Cohort 4, Colorectal | Part B, Cohort Expansion - Cohort 5, Basket
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/6 | 1/8 | 0/7 | 0/8 | 1/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/3 | 0/6 | 8/8 | 2/7 | 5/8 | 5/9 | 2/8
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 5/6 | 8/8 | 6/7 | 8/8 | 9/9 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Dose Escalation - OBI-888 5 mg/kg (N=5) | Part A, Dose Escalation - OBI-888 10 mg/kg (N=3) | Part A, Dose Escalation - OBI-888 20 mg/kg (N=6) | Part B, Cohort Expansion - Cohort 1, Pancreatic (N=8) | Part B, Cohort Expansion - Cohort 2, Esophageal (N=7) | Part B, Cohort Expansion - Cohort 3, Gastric (N=8) | Part B, Cohort Expansion - Cohort 4, Colorectal (N=9) | Part B, Cohort Expansion - Cohort 5, Basket (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Dose Escalation - OBI-888 5 mg/kg (N=5) | Part A, Dose Escalation - OBI-888 10 mg/kg (N=3) | Part A, Dose Escalation - OBI-888 20 mg/kg (N=6) | Part B, Cohort Expansion - Cohort 1, Pancreatic (N=8) | Part B, Cohort Expansion - Cohort 2, Esophageal (N=7) | Part B, Cohort Expansion - Cohort 3, Gastric (N=8) | Part B, Cohort Expansion - Cohort 4, Colorectal (N=9) | Part B, Cohort Expansion - Cohort 5, Basket (N=8)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 3 (3) | 3 (6) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (6) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Fatigue (General disorders) | 2 (2) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 2 (3) | 3 (4)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 | 1 | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (8) | 2 (4) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT03573544/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT03573544/SAP_001.pdf